CLINICAL TRIAL: NCT04406584
Title: Intranasal Injection of Platelet-rich Plasma Versus Saline for Treatment of Olfactory Dysfunction
Brief Title: Intranasal Injection of PRP Versus Saline for Treatment of Olfactory Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Zara M. Patel, Professor and Director of Endoscopic Skull Base Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-55353
Record Dates: First submitted 2020-05-11; First posted 2020-05-28 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Olfactory Disorder; Olfaction Disorders; Olfactory Nerve Injuries; Olfactory Nerve Disorder; Olfactory Nerve Diseases; Covid19; Post-Viral Disorder
Keywords: olfactory; olfactory loss; anosmia; hyposmia; olfactory dysfunction; prp; platelet enriched plasma; platelet rich plasma; endoscopic; covid19; post-viral disorder
MeSH Terms: conditions — Olfaction Disorders; Olfactory Nerve Injuries; Olfactory Nerve Diseases; COVID-19; Anosmia; Insomnia, Fatal Familial

STUDY DESIGN:
Intervention Model Description: Comparison of two randomized groups
Who Masked: Participant
Masking Description: Blindfold during injection and during portions of the smell test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): Injection of 1cc saline into olfactory cleft x4
  Interventions: Procedure: Injection into olfactory cleft
- Platelet Rich Plasma (Experimental): Injection of 1cc patient's own platelet rich plasma (PRP) into olfactory cleft x4
  Interventions: Procedure: Injection into olfactory cleft

INTERVENTIONS:
Procedure: Injection into olfactory cleft — Already stated above.

SUMMARY:
This randomized clinical trial will evaluate the benefit of platelet-rich plasma (PrP) in the treatment of olfactory dysfunction. PrP can be isolated from a patient's own blood and has been found in previous studies to have anti-inflammatory and pro-regenerative properties. It has been used across multiple specialties, such as Orthopedics, Facial Plastics, Dermatology, Neurology in injected form to treat a wide variety of tissues to encourage the body's inherent regenerative capacity. The investigators have completed a pilot study here evaluating it's use in olfactory loss which demonstrated safety and also suggested efficacy. Therefore, the investigators aim to assess the ability of PrP to improve olfactory function in patients with decreased sense of smell.

DETAILED DESCRIPTION:
Olfactory dysfunction constitutes a common impairment in the general population, affecting nearly 20 million in the USA and severely impairing quality of life. Unfortunately, this problem is often permanent, and no effective treatment is available at this time. Although many etiologies exist for olfactory loss, the underlying pathology is thought to be permanent damage to the olfactory bulb, nerves or basal cells of the olfactory system. Platelet-rich plasma (PRP) is an autologous treatment derived from a patient's own blood and has been found to have pro-nerve regenerative properties in animal and human studies. A small pilot study at the principal investigator's institution demonstrated improved olfactory thresholds in patients with partial olfactory loss who received PrP injections. In this randomized clinical trial, the investigators aim to further evaluate the ability of PRP injections to restore olfactory function in human subjects. Given the lack of effective current treatments, a therapeutic benefit of PrP would represent a crucial advancement in research and treatment of olfactory loss, which affects a large swath of the population.

Patients will be seen at the Stanford Sinus center, or at the newly added collaborating institution UCSD, and those with smell loss will be identified by the clinically validated patient directed survey: The UPSIT (University of Pennsylvania Smell Identification Test). They will undergo nasal endoscopy to exclude structural causes of smell loss including mass or tumor. Nasal endoscopy will be performed to exclude structural causes of olfactory, using topical anesthesia (1% phenylephrine & 4% lidocaine topical spray). THESE ABOVE STEPS CONSTITUTE STANDARD OF CARE FOR EVALUATION OF OLFACTORY LOSS.

The timing of the initial research visit will depend on the evolution of the current covid-19 pandemic and adhere to Stanford guidelines regarding research visits. At the initial research visit, patients meeting inclusion criteria will be evaluated in a procedure room at the Stanford Sinus center. A baseline Sniffin' sticks smell test will be performed (see below). A small vial of blood will be drawn from the patient at the Blake Wilbur first floor laboratory. The research coordinator will walk the patient back to clinic along with the patient's blood smple. PRP will be isolated from the blood by the study investigator, following manufacturer instructions from the PurePRP preparation kit (Emcyte corporation), which will involve use of a centrifuge located in the clinic for this purpose. 0.5 mL of the PRP solution will be set aside for platelet quantification. From the remaining PRP solution, patients will then receive 1ml of autologous PrP or sterile saline (0.9% Sodium Chloride), which will be injected into the superior septum mucosa near the olfactory groove bilaterally. Patients will be blindfolded during injection to prevent identification of the injected specimen, and will previously be randomized in a 1:1 ratio via a random number generator. Patients will be monitored for side effects for 15 minutes. (We routinely perform nasal endoscopy with injection and associated procedures in our clinic, which patients tolerate very well.) Injections will then be performed twice more at 2-weeks and 4-weeks after the initial injection, for a total of 3 biweekly injections. ALL OF THE ABOVE STEPS ARE FOR RESEARCH PURPOSES.

The Sniffin' Sticks test is a validated, non-invasive assessment of olfactory function via presentation of scented felt pens to blindfolded patients. The output is the TDI score (threshold, discrimination, identification). The TDI score will be recorded at baseline (initial research visit), and then at 1-month and 3-months after the initial test, for a total of 3 tests. The first test will occur before the first injection, and the second test will be performed before the third injection. There will be no injection at the last (third) test. THE ABOVE VISITS ARE FOR RESEARCH PURPOSES.

The study time-line is summarized as follows Visit 1: 1st Sniffin' Sticks test, 1st injection Visit 2: 2 weeks after Visit 1, second injection Visit 3: 4 weeks after Visit 1, second test, third injection Visit 4: 3 months after Visit 1, third test

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age
* Patients who have olfactory loss (based off of UPSIT score <= 33 out of 40)
* Patients who also have an age-adjusted TDI Sniffin' Sticks score that demonstrates hyposmia (TDI>16 and <30)
* Etiology of olfactory loss is due to URI or idiopathic
* At least 6 months of olfactory loss but less than 12 months
* Patients can have been previously treated with oral and topical steroids but this is not a requirement
* Patients will receive concurrent olfactory training - the practice of smelling strong odors (standard of care)
* Be able to read and understand English
* Agree to participate in the study
* Be able and willing to provide Informed Consent

Exclusion Criteria:

* Patients < 18 years of age
* Pregnant females
* Patient who have any structural abnormalities on nasal endoscopy or radiographic imaging
* Olfactory loss due to trauma, chronic sinusitis / inflammation / polyps, neoplasms, or neurodegenerative diseases
* Patients who have had olfactory loss > 12 months
* Patients with bleeding disorders or on blood thinners such as coumadin and plavix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Smelling ability | 6 months
  Using Sniffin' Sticks olfactory testing pens to test smell

CONTACTS AND LOCATIONS:
Overall Officials: Zara M. Patel, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California - San Diego, San Diego, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan CH, Mundy DC, Patel ZM. The use of platelet-rich plasma in treatment of olfactory dysfunction: A pilot study. Laryngoscope Investig Otolaryngol. 2020 Feb 21;5(2):187-193. doi: 10.1002/lio2.357. eCollection 2020 Apr. PMID 32337347
- [Result] Yan CH, Jang SS, Lin HC, Ma Y, Khanwalkar AR, Thai A, Patel ZM. Use of platelet-rich plasma for COVID-19-related olfactory loss: a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Jun;13(6):989-997. doi: 10.1002/alr.23116. Epub 2022 Dec 21. PMID 36507615
- See also: Dr. Patel's Stanford University School of Medicine Profile and Link to Donate to Research — https://profiles.stanford.edu/zara-patel